CLINICAL TRIAL: NCT07245446
Title: A Phase II Clinical Study of Ivonescimab Combination Therapy as First-Line Treatment for Extensive-Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: A Study of Ivonescimab in First-Line ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-214
Record Dates: First submitted 2025-09-29; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ivonescimab + AK117 + Chemotherapy (Experimental)
  Interventions: Drug: Ivonescimab; Drug: AK117; Drug: Etoposide; Drug: Carboplatin (AUC 5)
- Ivonescimab + Cadonilimab + Chemotherapy (Experimental)
  Interventions: Drug: Ivonescimab; Drug: Cadonilimab; Drug: Etoposide; Drug: Carboplatin (AUC 5)
- Ivonescimab + Chemotherapy (Experimental)
  Interventions: Drug: Ivonescimab; Drug: Etoposide; Drug: Carboplatin (AUC 5)

INTERVENTIONS:
Drug: Ivonescimab — Administered intravenously at a specified dose and frequency.
Drug: Cadonilimab — Administered intravenously at a specified dose and frequency.
  Arms: Ivonescimab + Cadonilimab + Chemotherapy
Drug: AK117 — Administered intravenously at a specified dose and frequency.
  Arms: Ivonescimab + AK117 + Chemotherapy
Drug: Etoposide — Administered intravenously at 100 mg/m² on Days 1-3 of each 3-week cycle for 4 cycles.
Drug: Carboplatin (AUC 5) — Administered intravenously at AUC 5 on Day 1 of each 3-week cycle for 4 cycles.

SUMMARY:
The goal of this clinical trial is to learn if different combinations of a drug called Ivonescimab, along with chemotherapy and other investigational drugs, are safe and effective for the initial treatment of adults with extensive-stage small cell lung cancer (ES-SCLC).

The main questions the study aims to answer are:

* What side effects do participants experience from these combination treatments?
* How well do the treatments work to shrink tumors?

Researchers will compare three groups to see which combination works best. All participants will receive Ivonescimab and chemotherapy (etoposide and carboplatin). The differences are:

* Group 1 will also receive an additional drug called AK117.
* Group 2 will also receive a different additional drug called Cadonilimab.
* Group 3 will receive Ivonescimab and chemotherapy only.

Participants will:

* Be assigned by chance to one of the three groups.
* Undergo an initial treatment phase (about 3 months), receiving chemotherapy plus the specific study drugs for their group.
* If the treatment is effective and side effects are manageable, continue with a maintenance phase using only the study drugs (without chemotherapy) for up to 2 years.
* Attend regular clinic visits for check-ups, blood tests, and imaging scans (like CT scans) to see how they are responding to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC).
* No prior systemic therapy for ES-SCLC.
* At least one measurable lesion as defined by RECIST v1.1.
* Age 18 to 75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function.

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastases (Treated, stable brain metastases are allowed).
* History of severe hypersensitivity to monoclonal antibodies.
* Active autoimmune disease requiring systemic treatment within the past 2 years.
* Significant cardiovascular disease.
* Active hepatitis B or C, or HIV infection.
* Interstitial lung disease or non-infectious pneumonitis.
* Significant bleeding tendency or risk, including tumor invasion of major blood vessels.
* Pregnancy or lactation.
* Other active malignancies within 5 years prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years.
  The proportion of participants achieving a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR), as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Incidence of Adverse Events (AEs) | From first dose up to 90 days after last dose.
  The number and percentage of participants experiencing any Adverse Event (AE). An AE is defined as any untoward medical occurrence in a participant administered a study drug, which may not have a causal relationship with the treatment. Severity will be graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 2 years.
  The proportion of participants achieving a BOR of CR, PR, or Stable Disease (SD), as assessed by the investigator per RECIST v1.1.
Duration of Response (DoR) | Up to approximately 2 years.
  For responders (participants achieving CR or PR), DoR is defined as the time from the first documented evidence of CR or PR until the first documented disease progression or death from any cause, whichever occurs first, per RECIST v1.1.
Time to Response (TTR) | Up to approximately 2 years.
  For responders (participants achieving CR or PR), TTR is defined as the time from the start of study treatment to the first documented objective response (CR or PR), per RECIST v1.1.
Progression-Free Survival (PFS) | Up to approximately 2 years.
  PFS is defined as the time from the start of study treatment to the first documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 5 years.
  OS is defined as the time from the start of study treatment to death from any cause.
Serum concentrations of Ivonescimab, Cadonilimab, and AK117 | Up to approximately 2 years.
  Serum concentrations of Ivonescimab, Cadonilimab, and AK117 will be measured to characterize the pharmacokinetic (PK) profiles.
Incidence of Anti-drug Antibodies (ADA) | Up to approximately 2 years.
  The immunogenicity will be assessed by the incidence of participants who develop detectable anti-drug antibodies (ADA) against Ivonescimab, Cadonilimab, and/or AK117.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Pulmonary Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No